CLINICAL TRIAL: NCT03711942
Title: Comparison of Healing of Apical Periodontitis in Periodontally Diseased and Healthy Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Gaurav Endo
Record Dates: First submitted 2018-10-11; First posted 2018-10-19 (Actual); Last update posted 2018-10-19 (Actual); Status verified 2018-10

CONDITIONS: Apical Periodontitis
Keywords: Root canal treatment, intraorifice barrier.
MeSH Terms: conditions — Periapical Periodontitis | interventions — Alkalies

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Periodontally Healthy IOB (Active Comparator): Intra orifice barrier (IOB) was placed in periodontally healthy molar.
  Interventions: Procedure: Intra orifice barrier
- Periodontally Healthy Base (Experimental): 2mm thick base was applied in periodontally health teeth.
  Interventions: Procedure: Base
- Periodontally healthy control (Experimental): coronal access was restored with composite resin without any base.
  Interventions: Procedure: Control
- Periodontally diseased IOB (Active Comparator): Intra orifice barrier (IOB) was placed in periodontally healthy molar
  Interventions: Procedure: Intra orifice barrier
- Periodontally diseased Base (Active Comparator): 2mm thick Base of GIC was applied under composite restoration
  Interventions: Procedure: Base
- Periodontally diseased control (Active Comparator): coronal access was restored with composite resin without any base
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: Intra orifice barrier — After primary root canal treatment, Glass Ionomer Cement (KetacTM Molar, 3M ESPE) applied as intraorifice barrier 3mm inside canal from root canal orifice in first group, as 2mm base on floor of pulp chamber in second group and direct composite restoration in 3rd group without Intraorifice barrier or base.3mm GP in the orifice was removed and intraorifice barrier and 2mm thick base was given of GIC.
  Arms: Periodontally Healthy IOB; Periodontally diseased IOB
Procedure: Base — After primary root canal treatment, Glass Ionomer Cement (KetacTM Molar, 3M ESPE) applied as intraorifice barrier 3mm inside canal from root canal orifice in first group, as 2mm base on floor of pulp chamber in second group and direct composite restoration in 3rd group without Intraorifice barrier or base.2mm thick Base of GIC was applied over the orifice before composite restoration
  Arms: Periodontally Healthy Base; Periodontally diseased Base
Procedure: Control — After primary root canal treatment, Glass Ionomer Cement (KetacTM Molar, 3M ESPE) applied as intraorifice barrier 3mm inside canal from root canal orifice in first group, as 2mm base on floor of pulp chamber in second group and direct composite restoration in 3rd group without Intraorifice barrier or base.coronal accees upto orifice was restored with composite resin
  Arms: Periodontally diseased control; Periodontally healthy control

SUMMARY:
Periodontal health may jeopardize the success of endodontic treatment.Intraorifice barrier apart from enhancing probability of success of endodontic treatment may also augment periodontal therapy as intra pulpal infection is known to contribute in worsening of periodontal health by promoting marginal bone loss and pocket formation.This study compared the apical healing in healthy and periodontally compromised teeth and evaluated the effect of intra orifice barrier and base in the healing of apical periodontitis.

DETAILED DESCRIPTION:
Endodontic treatment comprises bio-mechanical preparation of root canal system, chemical debridement and obturation with inert material. Various prognostic factors like adequacy of root filling, pre-operative size of periapical lesion on radiograph, type and location of teeth, periodontal status of the teeth and coronal restoration may play role in the success of endodontic treatment.

In the presence of defective coronal seal percolation of saliva and microbes may take place causing treatment failure. This assumption has acquired support mainly from various in-vitro studies which has demonstrated penetration of dye /microbe / radioactive tracer along root filling. Marshall and Massler in an in-vitro study using radioisotopes were first to highlight effect of coronal leakage and later Swanson and Madison in a study involving 70 extracted single rooted human teeth showed complete dye penetration throughout obturation material and along the canal walls. Since then there has been a renewed interest in the endodontic community in exploring relation of coronal seal with prognosis of endodontic treatment.

In a retrospective study Ray and Trope concluded that coronal restoration has greater impact on success of endodontic therapy rather than quality of root filling. However, various other epidemiological studies failed to replicate this result. A recent meta-analysis stated that problem of coronal leakage may not be of that clinical significance as demonstrated in various in-vitro studies, though importance of good coronal restoration and good root filling in the success of endodontic treatment can't be denied.

Placing an additional protective barrier in the coronal portion of the root canal has been recommended to minimize microleakage and facilitate healing of apical periodontitis. Intraorifice barrier apart from enhancing probability of success of endodontic treatment may also augment periodontal therapy as intra pulpal infection may also contribute in worsening of periodontal health by promoting marginal bone loss and pocket formation. Similarity between microflora of periodontium and root canal has led to a view that the communication between the two exists, and can potentially affect status of one another. The observations on this issue have been conflicting in nature with some authors reporting pulpal necrosis due to periodontal disease, and others reporting normal teeth regardless of severity of periodontal disease (Zehnder). Stassen et al. in a retrospective study observed more signs of apical periodontitis in teeth with reduced marginal support. They also reported significant influence of coronal extent of obturation on outcome of endodontic treatment in periodontally compromised patients. Significantly less incidence of apical periodontitis was seen where gutta percha was apical to marginal bone as compared to gutta percha being coronal to marginal bone. It is evident that the interrelationship between root canal and periodontium is complicated, and still not fully understood on account of lack of studies exploring the topic So far no prospective clinical trial has investigated the effect of periodontal status on healing of apical periodontitis. Also in absence of a clinical study substantial amount of doubt still persists whether intraorifice barrier can emerge as an effective mean to prevent microleakage in furcation and root canals of a multirooted tooth which because of its anatomical aberrations poses stiff challenge for clinicians. Therefore aim of this study was to determine effect of the periodontal status on periapical healing and to determine effect of intracanal glass ionomer restoration as intraorifice barrier on treatment outcome of apical periodontitis.

Clinical procedure:

After initial periodontal therapy, Standard root canal treatment was done using standard protocol. The canals were prepared with Revo S instrument according to manufacturer instructions and obturation was done using gutta percha. First of all, local anesthesia was administered using 2% lignocaine hydrochloride with epinephrine 1:80,000 (ICPA Health Products Ltd, Ankleshwar, India) and tooth was isolated under rubber dam. Caries excavation was done and access cavity was prepared using carbide burs in high speed hand-piece with copious irrigation. The pulp chamber was debrided and all canal orifices were identified and coronally enlarged with low speed Gates Glidden drills (Mani Inc, Utsunomiya, Tochigi, Japan). Working length was determined using Root ZX apex locator (J. Morita, Irvine, CA) and verified radiographically. After creating glide path with #15 k-file, Revo-S (Micro Mega, Besancon, France) instruments were used in sequence as suggested by manufacturer with a rotational speed of 350 rpm at torque setting of 2.5 Ncm in gentle in-out motion. Irrigation was carried out using 5 mL of a 5.25% Sodium hypochlorite (NaOCl; PrevestDenpro Ltd, Jammu, India) solution between files with 26 gauge side vented needle (Neelkanth Healthcare Pvt. Ltd, Jodhpur, Rajasthan, India). After preparation, the root canals were irrigated with 5 mL 17% EDTA (Canallarge, Ammdent, Mohali, India) for 1 minute to remove smear layer, followed by final irrigation with 5 mL 5.25% NaOCl. The root canal was then dried using paper points and filled with laterally condensed gutta-percha (Meta Biomed Co Ltd, Korea) and zinc oxide eugenol sealer (Dental Products of India Ltd, New Delhi, India). Gutta-percha was cut with a heated instrument and vertically condensed right at the orifice opening of the canals.

The teeth were then randomly sub-divided into 3 experimental groups IOB, Base and Control. In IOB group gutta-percha was removed 3 mm from the coronal portion of the canal with heated plugger, while it was left at the level of orifice in base and control groups. Thereafter, coronal restoration of composite resin was done in all groups. In IOB group orifice was sealed with GIC and base of GIC was applied in both IOB and base group before composite restoration

ELIGIBILITY:
Inclusion Criteria:

* Permanent mandibular molar with pulpal necrosis as confirmed by negative response to pulp sensibility test (cold and electric pulp test),
* Radiographic evidence of apical periodontitis in the form of periapical radiolucency (minimum size ≥ 2 mm ~ 2 mm),
* Probing Depth of not more than 5mm.

Exclusion Criteria:

* Patient with diabetes,
* History of antibiotic intake in past 1 month,
* Presence of any immunocompromised conditions,
* Pregnant women, and
* Root filled and unrestorable teeth

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-10-15 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Healing of apical periodontitis | Baseline to one year
  Clinical success as depicted by absence of signs and symptoms, and radiographic success demonstrated by absence of periapical alterations (radiolucency at furcal or periapical region).

SECONDARY OUTCOMES:
Healing of marginal periodontitis | Baseline to one year
  improvement of periodontal parameters like probing depth (in millimeter) and marginal bone height (in millimeter).

IPD SHARING:
Plan to Share IPD: No